CLINICAL TRIAL: NCT01478711
Title: Comprehensive Clinical Decision Support (CDS) for the Primary Care of Premature Infants
Acronym: PreemieCDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-007241; 1RC1LM010471-01 (NIH)
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): A clinical decision support tool for the care and management of premature infants will be embedded into the electronic health record.
  Interventions: Other: Clinical Decision Support Tool
- No Intervention (No Intervention): No intervention, No clinical decision support tool will be used for non-intervention sites.

INTERVENTIONS:
Other: Clinical Decision Support Tool — A clinical decision support tool embedded within Epic will appear for children with a history of prematurity at the intervention sites.
  Arms: Intervention

SUMMARY:
This study will use a rules-based expert system embedded in an electronic health record (EHR) to extract, interpret, and present salient facts and recommendations related to the healthcare of premature infants.

DETAILED DESCRIPTION:
Premature infants are a vulnerable population with multiple inter-related health problems that put them at risk for poor outcomes. Electronic health records capture large amounts of information that may help guide decisions, but existing alert and reminder-based clinical decision support (CDS) frameworks do not adequately apply multiple overlapping care guidelines to complex patient histories to produce coherent clinical recommendations.

The primary objective of the study is to design and evaluate the usability of a CDS intervention to improve the quality of primary care for low birth weight (LBW) and very low birth weight (VLBW) premature infants from the time of intensive care nursery discharge through 24 months corrected gestational age

ELIGIBILITY:
Inclusion Criteria:

* All clinicians from participating practices.
* Premature Infants: Receive preventive healthcare from a participating practice at least twice during the study period; (2) age less than 24 months; and (3) birth weight less than 2000 g or gestational age at birth less than 35 weeks.

Exclusion Criteria:

-Residents will not eligible to participate in this study due to the fact that they receive significant ongoing education related to the inpatient and outpatient management of premature infants as part of their day-to-day training.

Ages: 20 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1517 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Evaluate usability of the intervention | 12 months
  Design and evaluation of the pre-implementation data-mining and expert system will employ usability methods from the human-computer interaction (HCI) field. The methods are based on the collection of quantitative and qualitative data where each method has specific metric-based goals that are to be achieved before the next phase. 10-20 clinicians, including attending physicians, nurse practitioners and nurses, from a single practice will be recruited to participate in the Usability Study.

SECONDARY OUTCOMES:
Evaluate effect on care process | 12 months
  The clinical decision support (CDS) intervention will be tested for correctness and usability prior to implementation. The effect on care processes will examine process outcomes in the following domains: (1) neonatal summary documentation; (2) growth and nutrition; (3) ophthalmology; (4) hearing, speech, and language; (5) development; (6) gastro-esophageal reflux; (7) broncho-pulmonary dysplasia; and (8) apnea of prematurity. The primary evaluation will examine the change in prevalence of these process outcomes between a 12 month pre-intervention phase and a 12 month intervention phase for bo

CONTACTS AND LOCATIONS:
Overall Officials: Robert Grundmeier, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital pf Philadelphia, Philadelphia, Pennsylvania, United States